CLINICAL TRIAL: NCT02911012
Title: Multiple Algorithms System Of All Scores in Embolism - MOSE
Brief Title: Multiple Algorithms System Of All Scores in Embolism (MOSE)
Acronym: MOSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Prof. Stefano de Franciscis, Full Professor of Surgery, University Magna Graecia
Other Study IDs: ER.ALL.2016.01
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Venous Thromboembolism; Risk Assessment; Risk Management
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: The identified population will be assessed on VTE risk according to the risk score PADUA, CAPRINI, KHORANA, and IMPROVE for BLD risk.

SUMMARY:
The aim of this study is to overcome the current limits of the scoring systems used to predict both the thrombotic (VTE) and hemorrhagic (BLD) risk for the patient. The main problem of these scoring systems is due to the high rigidity related to the score assigned at each risk item. The presence of an item assigns the full score for that item, without the possibility to moderate that item's score. The final class of risk, for the patient, is the sum of the scores of the selected items. The approach used for the assessment is based on the presence or absence of certain items that will be summed.

Starting from scoring system currently used for VTE (PADUA, CAPRINI, KHORANA) and also for BLD (IMPROVE), we will integrate all common items in a single scoring system managed by risk management algorithms that can identify the different classes of risk.

DETAILED DESCRIPTION:
The term venous thromboembolism is used to define any thrombotic event within the venous system with or without pulmonary embolism (PE). Deep vein thrombosis (DVT) is still, together with PE, possibly resulting therefrom, one of the most common and serious complications that may occur in specific risk patients.

The current diagnostic systems allow to verify the presence, more quickly and frequently of DVT; moreover, DVT and PE if not promptly diagnosed determine the underestimation of their true incidence with negative consequences on morbidity and mortality.

The proposed systems also can be particularly incisive in monitoring the recurrence risk of thromboembolic disease, that currently is entrusted exclusively to biological predictive diagnostics (d-dimer, etc.) or diagnostic imaging (ultrasound, angio-ct etc.). These monitoring methodologies were often burdened by an excess of false positives and, in any case, present not always affordable cost for the health system.

The innovative system is proposed as monitoring and risk management tool through simple repetition of the assessment.

VTE is the third leading cause of cardiovascular death after heart attack and stroke and in Italy the estimate is 100 new cases per year per 100,000 inhabitants. The VTE risk criteria are currently shared in the scientific community through the use of thrombotic risk tables generally accepted and validated like PADUA, CAPRINI, KHORANA, etc.

The score calculated puts the patient in a band of risk (low / medium / high) indicated by a number obtained by the sum of the detected risk factors. The identification of the risk level VTE (low / medium / high) involves the administration of therapy (antiplatelet and / or anticoagulant) according to the ACCP (American College of Chest Physicians' 2016).

Over the past years several scoring systems have been proposed. These systems are designed to stratify the risk of thrombosis in patients characterized by significant differences. In particular, some score systems consider risk factors not taken into account by others and some are applied to patient populations that present a high risk of VTE already known.

The risk score assessment in a patient cannot be based only on measurements of the binary questions (e.g. true or false) or using strict criteria in the analysis of physiological variables; this involves the possibility of incurring errors of evaluation, especially in those cases in which the patient manifests a borderline situation between a real risk and a situation of relative normality.

MOSE proposes an innovative approach to identify a multi-risk, both VTE and BLD, that take into account a series of variables, and situation, that the current score systems can't describe.

The proposed study want to test a system that supports the physician like a DSS (Decision Support System) in choosing the best therapy, to prevent VTE event, for the patient. Also, the study want to evaluate the actual role of risk factors in determining the VTE.

The system is suitable for further developments in the study of bleeding risk in patients with VTE risk and in the study of both risks (VTE vs BLD) as a function of time and therapies.

The study is retrospective and provides analysis of an outpatient population of general practitioner for a total of 15208 patients. To be eligible, the patients had to present at the doctor's office for a consultation related to a health disorder and to meet the following inclusion criteria: age ≥ 18 years, cooperative attitude, and signature of the informed consent form granting permission to use their personal health data.

The identified population will be assessed on VTE risk according to the risk score PADUA, CAPRINI, KHORANA, and IMPROVE for BLD risk.

The aim of this study is to implement a predictive system, based on fuzzy logic, capable to identify patients with the risk to develop a VTE event.

In the first part of the study the presence or absence of VTE events will be hidden at the researchers.

After calculating the MOSE risk score, results will be crossed with patients who actually had a VTE event, and then the results will be compared with the scores systems used in the study (PADUA, CAPRINI, KHORANA).

ELIGIBILITY:
Inclusion Criteria:

* the patients had to present at the doctor's office for a consultation related to a health disorder;
* age ≥ 18 years;
* cooperative attitude;
* signature of the informed consent form granting permission to use their personal health data;

Exclusion Criteria:

- patients not signing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is retrospective and provides analysis of an outpatient population of general practitioner for a total of 15208 patients
Sampling Method: Non-Probability Sample
Enrollment: 15208 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
VTE evaluation | 6 months
  After calculating the MOSE risk score, results will be crossed with patients who actually had a VTE event, and then the results will be compared with the scores systems used in the study (PADUA, CAPRINI, KHORANA)

SECONDARY OUTCOMES:
BLD evaluation | 6 months
  After calculating the MOSE risk score for BLD, results will be crossed with patients who actually had a bleeding risk, and then the results will be compared with the scores systems used in the study (IMPROVE).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano de Franciscis, M.D., Principal Investigator — University Magna Graecia of Catanzaro; Raffaele Serra, M.D., PhD., Study Chair — University Magna Graecia of Catanzaro; Matteo Di Minno, M.D., PhD, Study Chair — Federico II University
Locations (2):
- Italy (2):
  - University Magna Graecia of Catanzaro, Catanzaro
  - University Federico II of Naples, Naples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geerts WH, Pineo GF, Heit JA, Bergqvist D, Lassen MR, Colwell CW, Ray JG. Prevention of venous thromboembolism: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):338S-400S. doi: 10.1378/chest.126.3_suppl.338S. PMID 15383478
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Barbar S, Noventa F, Rossetto V, Ferrari A, Brandolin B, Perlati M, De Bon E, Tormene D, Pagnan A, Prandoni P. A risk assessment model for the identification of hospitalized medical patients at risk for venous thromboembolism: the Padua Prediction Score. J Thromb Haemost. 2010 Nov;8(11):2450-7. doi: 10.1111/j.1538-7836.2010.04044.x. PMID 20738765
- [Background] Obi AT, Pannucci CJ, Nackashi A, Abdullah N, Alvarez R, Bahl V, Wakefield TW, Henke PK. Validation of the Caprini Venous Thromboembolism Risk Assessment Model in Critically Ill Surgical Patients. JAMA Surg. 2015 Oct;150(10):941-8. doi: 10.1001/jamasurg.2015.1841. PMID 26288124
- [Background] Khorana AA, Kuderer NM, Culakova E, Lyman GH, Francis CW. Development and validation of a predictive model for chemotherapy-associated thrombosis. Blood. 2008 May 15;111(10):4902-7. doi: 10.1182/blood-2007-10-116327. Epub 2008 Jan 23. PMID 18216292
- [Background] de Franciscis S, Fregola S, Gallo A, Argiro G, Barbetta A, Buffone G, Calio FG, De Caridi G, Amato B, Serra R. PredyCLU: a prediction system for chronic leg ulcers based on fuzzy logic; part I - exploring the venous side. Int Wound J. 2016 Dec;13(6):1349-1353. doi: 10.1111/iwj.12529. Epub 2015 Nov 6. PMID 26542425